CLINICAL TRIAL: NCT01495988
Title: Randomized Phase II Trial of Vemurafenib (PLX4032/RG7204)/Cobimetinib (GDC-0973) With or Without Bevacizumab in Patients With Stage IV BRAFV600 Mutant Melanoma
Brief Title: Trial of Vemurafenib/Cobimetinib With or Without Bevacizumab in Patients With Stage IV BRAFV600 Mutant Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual; toxicity; change in priorities
Sponsor: Melanoma Research Foundation Breakthrough Consortium (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML27894; GEN-01 (Other: MRFBC)
Record Dates: First submitted 2011-12-09; First posted 2011-12-21 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-09

CONDITIONS: Melanoma; Metastatic Melanoma
Keywords: Metastatic melanoma; BRAF-mutant; Stage IV melanoma; Vemurafenib; Bevacizumab; Cobimetinib
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; Bevacizumab; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vemurafenib/Cobimetinib (Active Comparator): Vemurafenib will be given at a dose of 960 mg, orally, 2X a day to all patients. Cobimetinib will be given at a dose of 60mg, orally, 1X a day to all patients for 21 days, then 7 days off, in a 28 day treatment cycle. Patients will be assessed for toxicity every 4 weeks and be restaged for tumor response/progression every 8 weeks until week 48, then every 12 weeks thereafter. Patients will be followed until disease progression.
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib
- Vemurafenib/Cobimetinib + Bevacizumab (Experimental): Vemurafenib will be given at a dose of 960 mg, orally, 2X a day to all patients. Cobimetinib will be given at a dose of 60mg, orally, 1X a day to all patients for 21 days, then 7 days off, in a 28 day treatment cycle. Bevacizumab will be administered at the MTD (determined by phase Ib safety lead-in), intravenously, every 2 weeks. Patients will be assessed for toxicity every 4 weeks and be restaged for tumor response/progression every 8 weeks until week 48, then every 12 weeks thereafter. Patients will be followed until disease progression.
  Interventions: Drug: Vemurafenib; Drug: Bevacizumab; Drug: Cobimetinib
- Vemurafenib (Active Comparator): Vemurafenib will be given at a dose of 960 mg p.o. BID to all patients. Patients will be assessed for toxicity every 3 or 6 weeks (depending on the specific toxicity) and be restaged for tumor response/progression every 6 weeks until week 48, then every 12 weeks thereafter. Patients will be followed until disease progression.
  Interventions: Drug: Vemurafenib
- Vemurafenib + Bevacizumab (Experimental): Vemurafenib will be given at a dose of 960 mg p.o. BID to all patients. Patients assigned to the combination arm will also receive bevacizumab 15 mg/kg every IV every 3 weeks. Patients will be assessed for toxicity every 3 or 6 weeks (depending on the specific toxicity) and be restaged for tumor response/progression every 6 weeks until week 48, then every 12 weeks thereafter. Patients will be followed until disease progression.
  Interventions: Drug: Vemurafenib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib will be given at a dose of 960 mg, orally, 2X a day to all patients until disease progression, intolerable toxicity, patient request for discontinuation, or study termination by the sponsor.
  Other Names: Zelboraf
Drug: Bevacizumab — Patients assigned to the combination arm will also receive bevacizumab at 15mg/kg, intravenously, every 3 weeks.
  Other Names: Avastin
  Arms: Vemurafenib + Bevacizumab; Vemurafenib/Cobimetinib + Bevacizumab
Drug: Cobimetinib — Cobimetinib will be given at a dose of 60mg, orally, 1X a day to all patients for 21 days, then 7 days off, in a 28 day treatment cycle.
  Other Names: GDC-0973
  Arms: Vemurafenib/Cobimetinib; Vemurafenib/Cobimetinib + Bevacizumab

SUMMARY:
This phase 2 clinical trial randomizes patients with BRAF mutant melanoma to either (1) standard of care (SOC) - BRAF inhibitor vemurafenib in combination with MEK inhibitor cobimetinib; or, (2) SOC plus bevacizumab, an anti-VEGF antibody that suppresses new blood vessel formation and can stimulate the immune system. Previous clinical studies in melanoma have shown that bevacizumab may improve clinical benefit (progression free survival) if combined with ipilimumab or abraxane. Preclinical studies suggest that VEGF increase plays a role in resistance to BRAF inhibitors. This randomized study will ask whether the addition of bevacizumab to targeted therapy SOC in BRAF mutant melanoma can improve response rates and clinical benefit. Patients may have received no therapy for advanced disease or up to 2 prior therapies, excluding BRAF and MEK inhibitors.

DETAILED DESCRIPTION:
In this study, the drugs being used are vemurafenib, cobimetinib, and bevacizumab. Vemurafenib has been approved by the FDA for treatment of patients with advanced melanoma that harbors a BRAF mutation. However, vemurafenib in combination with cobimetinib has not been approved by the FDA for the treatment of cancer. Bevacizumab has been approved by the FDA for use in combination with first line chemotherapies for treatment of patients with colorectal, breast and lung cancer. Bevacizumab has not been approved for use in patients with metastatic melanoma.

Vemurafenib and cobimetinib attack different proteins that cause cancer cells to grow. Vemurafenib works by blocking a protein called B-RAF. Researchers have found that a large number of melanomas have mutations (changes) in the BRAF gene. The BRAF gene codes for a protein called B-RAF, which is involved in sending signals in cells that can lead to cell growth. Research has determined that mutations in the BRAF gene at the V600 position cause a change in the B-RAF protein that can drive the growth and spread of melanoma cells. Vemurafenib works by preventing these altered B-RAF proteins from working, and thereby may block the growth and spread of cancer cells in patients with melanoma. Cobimetinib works by blocking a protein called MEK. MEK has been known to promote growth in cancer that carries either a mutation in the BRAF or KRAS genes. The vemurafenib/cobimetinib combination has been used in prior clinical studies. Information from those other research studies suggests that these drugs can shrink melanoma tumors in the majority of patients and slow tumor growth as compared to standard chemotherapy. Another drug to block the BRAF and MEK proteins was recently approved by the FDA in the treatment of patients with B-RAFV600 mutant melanoma. The researchers want to see if using vemurafenib and cobimetinib together will work in a similar way to treat malignant melanoma.

Bevacizumab is a humanized monoclonal antibody (a type of protein that is normally made by the immune system to help defend the body from infection and cancer) produced by using recombinant DNA technology. Bevacizumab is an antibody directed against vascular endothelial growth factor or VEGF. VEGF is a potent, specific growth factor with a well-defined role in normal and abnormal blood vessel formation. It is present in a wide variety of normal tissues, but is produced in excess by most solid cancers (tumors). In the setting of cancer, VEGF promotes the growth of blood vessels that bring nutrients to tumor cells. Its expression by the tumor has been associated with worse outcome in patients with a number of tumors types including melanoma. In laboratory experiments, bevacizumab inhibits the growth of several different types of human cancer cells by blocking the effects of VEGF.

The purpose of this research study is to determine the effectiveness of using the study drugs vemurafenib, cobimetinib, and bevacizumab together relative to vemurafenib and cobimetinib alone. This study will investigate whether using both study drugs lengthens the amount of time before participants' melanoma worsens, increases the number of people whose melanoma responds to treatment and what the side effects are of using the drugs together rather than separately.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histological or cytological confirmed melanoma that is metastatic or unresectable stage IIIc and clearly progressive.
2. Patients must have melanoma that is documented to contain a BRAFV600E or BRAFV600K mutation by a FDA-approved test.
3. Age >= 18 years.
4. Women must not be pregnant due to the fact that the effects of vemurafenib, cobimetinib, and/or bevacizumab on the developing human fetus are unknown. For this reason and because antiangiogenic agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence; defined in Appendix G) prior to study entry and for the duration of study participation. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately.
5. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
6. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with bevacizumab, cobimetinib, and vemurafenib, female participants who are breastfeeding must agree to discontinue nursing prior to Day 1 of the study.
7. Patients must have measurable disease as defined in Section 10.1 (cutaneous lesions measuring at least 1 cm will be considered measurable). Baseline CT or MRI scans of measurable disease sites must be performed within 4 weeks of study entry.
8. Patients must have discontinued immunotherapy or other systemic therapy including investigational agents at least 4 weeks prior to entering the study and have recovered from adverse events due to those agents. Patients must agree to not receive any other investigational agents during study participation.
9. Patients must have an ECOG performance status of 0, 1, or 2.
10. Patients must have the following baseline laboratory values:

    1. White Blood Count > 3,000/mm3
    2. Absolute Neutrophil Count > 1,500/mm3
    3. Platelet Count > 100,000/mm3
    4. Serum creatinine < 1.5 x upper limit of normal (ULN) or serum creatinine clearance (CrCl)> 40ml/min (CrCl= Wt (kg) x (140-age)*/72 x Cr. level, *female x 0.85)
    5. Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) < 3 x ULN (< 5 x ULN for patients with documented liver metastases)
    6. Alkaline Phosphatase =< 2 x ULN (=< 5 x ULN for patients with known liver involvement and =< 7 x ULN for patients with known bone involvement)
    7. International Normalized Ratio (INR) < 1.5 and aPTT within 1.1 x ULN
    8. Total Bilirubin < 1.5 x ULN
    9. UPC ratio < 1.0 at screening or 24 hours urine protein < 1 gm (Appendix D)
11. Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients may not have received more than 2 prior systemic treatment regimens for distant metastatic disease. The following prior therapy is permitted in either the adjuvant or metastatic disease setting, provided treatment is discontinued at least 4 weeks prior to initiating study treatment:

   1. Immunotherapy, such as interferon, interleukin-2, GM-CSF, ipilimumab, anti-PD1 or other experimental agent.
   2. Cytotoxic chemotherapy, such as dacarbazine, temozolomide, carboplatin +/-paclitaxel.
2. Patients may not have had radiation therapy within the last 4 weeks prior to initiation of study treatment.
3. Patients who have had prior VEGF pathway inhibitor, BRAF or MEK inhibitor therapy are ineligible.
4. Patients must have no clinical evidence of active brain metastasis. Patients with a history of brain metastases must meet all of the following criteria:

   1. Have completed treatment greater than 4 weeks prior to enrollment.
   2. Have CNS lesions that are confirmed to be stable or regressing on imaging since the time of the last CNS treatment including the pre-treatment CT or MRI scan for this trial.
   3. Patients must have no residual neurologic symptoms while taking no steroids, a stable or decreasing dose of steroids, or a stable dose of anti-seizure medication for the 2 weeks prior to enrollment.
5. Patients must not have other concurrent uncontrolled malignancies, defined as a malignancy that currently requires therapy or other intervention. Patients with suspected cuSCCs should have them excised prior to study registration. Surgical resection should not be performed within 7 days of starting protocol therapy.
6. Patients may not have had a major surgical procedure, open biopsy (excluding skin cancer resection, cutaneous/subcutaneous melanoma metastasis resection or biopsy or vascular access device insertion), or significant traumatic injury within 28 days prior to Day 1, or have an anticipated need for major surgical procedure or a planned elective surgical procedure during the course of the study.
7. Patients may not have had a core biopsy, skin cancer resection, or other minor surgical procedure, including placement of a vascular access device, within 7 days prior to Day 1 of the protocol.
8. Patients must not have a serious intercurrent illness including, but not limited to:

   1. Ongoing or active infection requiring parental antibiotics on Day 1
   2. A history of malabsorption or other condition that would interfere with absorption of vemurafenib or cobimetinib.
   3. History of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
   4. History of congenital long QT syndrome or mean corrected QTc interval > 450 msec at baseline
   5. Clinically significant cardiovascular disease, defined as any of the following conditions:

   i. Uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) ii. Prior history of hypertensive crisis or hypertensive encephalopathy iii. Myocardial infarction within 6 months iv. Unstable angina v. New York heart association grade II or greater congestive heart failure (Appendix C) vi. Serious cardiac arrhythmia requiring medication vii. LVEF < 50% or below institutional limit of normal f) History of stroke of TIAs within 6 months prior to Day 1 g) Grade II or greater peripheral vascular disease within 1 year prior to study entry or other significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1 h) Serious, non-healing wound, active ulcer, or untreated bone fracture i) History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1 j) Known hypersensitivity to any component of bevacizumab k) Known CNS disease, except for stable or regressing brain metastases. l) Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation) m) Psychiatric illness/social situations that would limit compliance with study requirements.

   n) Significant ocular issues including history of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, retinal vein occlusion (RVO), or neovascular macular degeneration. The risk factors for RVO are listed below. Patients should be excluded if they have the following conditions:
   1. Uncontrolled glaucoma with intra-ocular pressures >21mm Hg
   2. Serum cholesterol >= Grade 2
   3. Hypertriglyceridemia >= Grade 2
   4. Hyperglycemia (fasting) >= Grade 2
9. Patients must not have the following foods/ supplements at least 7 days prior to initiation of and during study treatment:

   1. St. John's wort or hyperforin (potent cytochrome P450 CYP3A4 enzyme inducer)
   2. Grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor).
10. Because patients with immune deficiency are at increased risk of lethal infections when treated with bone marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with bevacizumab, vemurafenib and cobimetinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Atkins, MD, Principal Investigator — Beth Israel Deaconess Medical Center; F. Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (14):
- United States (14):
  - The Angeles Clinic, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Harry and Jeannette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYU Clinical Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - OSU Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight subjects were randomized under protocol v2.0 with the first subject enrolled on 8/13/2013. Two subjects were enrolled under protocol v4.0 with the first subject enrolled on 6/19/2015. The study was permanently closed on 6/13/2016. All subjects were recruited from Melanoma Research Foundation Breakthrough Consortium (MRFBC) clinical sites.
Pre-assignment Details: Participants has to meet the eligibility criteria prior to enrollment into the study.
Groups:
- Vemurafenib/Cobimetinib: Vemurafenib: Vemurafenib will be given at a dose of 960 mg, orally, 2X a day to all patients until disease progression, intolerable toxicity, patient request for discontinuation, or study termination by the sponsor.
  Cobimetinib: Cobimetinib will be given at a dose of 60mg, orally, 1X a day to all patients for 21 days, then 7 days off, in a 28 day treatment cycle.
  Patients will be assessed for toxicity every 4 weeks and be restaged for tumor response/progression every 8 weeks until week 48, then every 12 weeks thereafter. Patients will be followed until disease progression.
- Vemurafenib/Cobimetinib + Bevacizumab: Vemurafenib: Vemurafenib will be given at a dose of 960 mg, orally, 2X a day to all patients until disease progression, intolerable toxicity, patient request for discontinuation, or study termination by the sponsor.
  Bevacizumab: Patients assigned to the combination arm will also receive bevacizumab at 15mg/kg, intravenously, every 3 weeks.
  Cobimetinib: Cobimetinib will be given at a dose of 60mg, orally, 1X a day to all patients for 21 days, then 7 days off, in a 28 day treatment cycle.
  Patients will be assessed for toxicity every 4 weeks and be restaged for tumor response/progression every 8 weeks until week 48, then every 12 weeks thereafter. Patients will be followed until disease progression.
- Vemurafenib: Vemurafenib will be given at a dose of 960 mg p.o. BID to all patients.
  Patients will be assessed for toxicity every 3 or 6 weeks (depending on the specific toxicity) and be restaged for tumor response/progression every 6 weeks until week 48, then every 12 weeks thereafter.
- Vemurafenib + Bevacizumab: Vemurafenib will be given at a dose of 960 mg p.o. BID to all patients.
  Patients assigned to the combination arm will also receive bevacizumab 15 mg/kg every IV every 3 weeks.
  Patients will be assessed for toxicity every 3 or 6 weeks (depending on the specific toxicity) and be restaged for tumor response/progression every 6 weeks until week 48, then every 12 weeks thereafter.
Period: Vem +/- Bev (Protocol v2.0)
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab
Started | 0 | 0 | 5 | 3
Completed | 0 | 0 | 5 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Vem/Cobi +/- Bev (Protocol v4.0)
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab
Started | 0 | 2 | 0 | 0
Completed | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab | Total
Number analyzed (Participants) | 0 | 2 | 5 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0 | 0 | 0
  Between 18 and 65 years |  | 0 | 1 | 3 | 4
  >=65 years |  | 2 | 4 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1 | 1 | 3
  Male |  | 1 | 4 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0 | 1 | 1
  Not Hispanic or Latino |  | 2 | 5 | 2 | 9
  Unknown or Not Reported |  | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 | 0 | 0
  Asian |  | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 | 0 | 0
  Black or African American |  | 0 | 0 | 0 | 0
  White |  | 2 | 5 | 3 | 10
  More than one race |  | 0 | 0 | 0 | 0
  Unknown or Not Reported |  | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States |  | 2 | 5 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: To establish the maximum tolerated dose (MTD) of bevacizumab in combination with vemurafenib and cobimetinib.
Time Frame: Until MTD determined (up to 6 months)
Population: The trial was terminated prematurely during the phase Ib safety lead-in and outcome measures were not analyzed. MTD could not be determined.
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Median Progression-free Survival
Description: To compare median progression-free survival (PFS) of patients with stage IV, BRAFV600E or BRAFV600K melanoma treated with vemurafenib/cobimetinib versus vemurafenib/cobimetinib and bevacizumab.
Time Frame: Time between randomization and disease progression (~10-15 months)
Population: The trial was terminated prematurely during the phase Ib safety lead-in and outcome measures were not analyzed due to significantly underpowered data and the MTD being undetermined.
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Overall Survival
Description: Compare overall survival (OS) of patients with stage IV, BRAFV600E/K melanoma treated with vemurafenib/cobimetinib versus vemurafenib/cobimetinib and bevacizumab.
Time Frame: Time between randomization and death due to any cause (overall survival rates also to be assessed at 12 and 18 months)
Population: as for outcome 2
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Response Rates
Description: Compare response rate (RR) of patients with stage IV, BRAFV600E/K melanoma treated with vemurafenib/cobimetinib versus vemurafenib/cobimetinib and bevacizumab.
Time Frame: From time of randomization to time of disease progression (restaging for tumor response to occur every 8 wks until wk 48, then every 12 wks thereafter)
Population: as for outcome 2
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Toxicity and Safety Profile
Description: Describe the toxicity and safety profile of treatment with vemurafenib/cobimetinib versus vemurafenib/cobimetinib and bevacizumab in patients with stage IV, BRAFV600E/K melanoma.
Time Frame: Until study completion
Population: as for outcome 2
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Effects of the Addition of Bevacizumab on Tumor Angiogenesis, Resistance Mechanisms and Immune Function
Description: Perform a variety of correlative studies aimed at understanding the effects of vemurafenib/cobimetinib, and bevacizumab administration relative to vemurafenib/cobimetinib on tumor angiogenesis, resistance mechanisms and immune function.
Time Frame: Upon completion of the protocol (3 years)
Population: The trial was terminated prematurely and outcome measures were not analyzed.
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Correlate Blood Markers of B-RAFV600 Mutation With Treatment Efficacy
Description: Assess the effectiveness of blood reverse transcription polymerase chain reaction (RT-PCR) assay for BRAFV600 as a surrogate biomarker for tumor response and resistance in patients receiving vemurafenib/cobimetinib +/- bevacizumab.
Time Frame: Upon completion of the protocol (3 years)
Population: as for outcome 2
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected from time of first study drug administration through 30 days following the last administration of study drug or study discontinuation/termination, whichever is earlier.
Description: Safety assessments will consist of monitoring and reporting the following adverse events (AEs):
  * Serious adverse events
  * Events that lead to drug discontinuation or interruption
  * All grade 3 and 4 toxicities
  * All deaths
  * Adverse events of special interest (AESI)
Arm/Group | Vemurafenib/Cobimetinib | Vemurafenib/Cobimetinib + Bevacizumab | Vemurafenib | Vemurafenib + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 0/0 | 1/2 | 5/5 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/0 | 2/2 | 3/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/0 | 2/2 | 4/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vemurafenib/Cobimetinib (N=0) | Vemurafenib/Cobimetinib + Bevacizumab (N=2) | Vemurafenib (N=5) | Vemurafenib + Bevacizumab (N=3)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated right femoral hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vemurafenib/Cobimetinib (N=0) | Vemurafenib/Cobimetinib + Bevacizumab (N=2) | Vemurafenib (N=5) | Vemurafenib + Bevacizumab (N=3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Incarcerated right femoral hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Development Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema Limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Unknown Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely on June 13, 2016. No further accrual to the study will occur.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No